CLINICAL TRIAL: NCT05509426
Title: Determining Who Benefits Most From Cognitive Rehabilitation for Attention and Memory in Multiple Sclerosis: A Randomised Controlled Feasibility Trial
Brief Title: Who Benefits Most From Cognitive Rehabilitation for Multiple Sclerosis?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: National Multiple Sclerosis Society (Other); University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21063
Record Dates: First submitted 2022-05-31; First posted 2022-08-22 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive an online cognitive rehabilitation programme, offered in addition to usual clinical care, to groups of 4-6 participants weekly for 10 sessions.
  Interventions: Behavioral: Cognitive Rehabilitation
- Usual Clinical Care (No Intervention): This group will receive only their usual clinical care, which may include information on cognitive problems as per clinical practice but not specific cognitive rehabilitation.

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — This cognitive rehabilitation will be tailored to each participant's cognitive status while maintaining a systematic treatment approach to attention and memory, following a study treatment manual. The intervention will include (i) restitution strategies to retain memory and attention functions including strategies to improve encoding and retrieval, (ii) compensation strategies, including internal mnemonics, use of external devices and ways of coping with attention and memory problems, (iii) the importance of errorless learning. The emphasis will be on identifying the most appropriate strategies to help individuals overcome their cognitive problems and in providing participants with a range of techniques, which they can adapt and use according to their needs. This is group based intervention that will take place remotely using MS Teams.
  Arms: Intervention Group

SUMMARY:
Over the last 20 years, there have been many studies investigating the efficacy of attention and memory rehabilitation for people with multiple sclerosis (MS) however, there appears to be a lack of conclusive evidence regarding the true effectiveness of this intervention. This could be because the participant samples recruited to these studies are often extremely varied in terms of socio-demographics and clinical characteristics, and it would be very unlikely that all people with MS would benefit from these interventions uniformly. Therefore, there is a need to explore which subgroups of people with MS benefit most from cognitive rehabilitation so that this information can be used to help clinicians and services make decisions as to whom this intervention is offered. Cognitive rehabilitation is not routinely provided on the NHS due to lack of resources. This research is important as it will allow these resources to be optimised and made available to those who need them, but also to allow clinicians to understand whether their patient is likely to benefit from cognitive rehabilitation before it is offered.

The primary aim of this study is to assess the feasibility and acceptability of undertaking a randomised controlled trial (RCT) to investigate the effectiveness of an online group-based cognitive rehabilitation programme with specific groups of people with MS. The secondary aim is to understand the impact that this intervention may have on various aspects of cognition such as memory, attention, and information processing. This will be assessed through various questionnaires and objective neuropsychological tests.

In addition, an algorithm has been developed following the secondary data analysis of a large RCT investigating group-based cognitive rehabilitation for people with MS. This algorithm may be able to determine who benefits most from cognitive rehabilitation, we will therefore use this as part of the data analysis to understand if the algorithm has the potential to be an accurate clinical prediction tool.

After completion of the cognitive rehabilitation, a small number of participants in the intervention group will be invited to take part in feedback interviews to give their views on the feasibility and acceptability of the group-based online cognitive rehabilitation and provide any suggestions for improvements for future trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 or over and under 70 years of age.
* Have MS, diagnosed at least 3 months prior to recruitment.
* Have cognitive deficits, defined as performance below the 25th percentile on the Brief Repeatable Battery of Neuropsychological Tests (BRBN).
* Able to speak English sufficiently to complete the cognitive assessments and take part in group sessions.
* Have access to laptop or PC that supports MS Teams.
* Able to give informed consent.

Exclusion Criteria:

* Vision or hearing problems, such that they are unable to complete the cognitive assessments, judged assessor.
* Have concurrent severe medical or psychiatric conditions which would prevent participants from engaging in treatment, if allocated.
* Are involved in other psychological intervention trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Acceptability and feasibility of conducting an online group-based cognitive rehabilitation programme. | Between the 3-month follow-up point and the 6-month follow-up point, up to 3 months.
  Feedback interviews will be conducted to understand the acceptability and feasibility of the intervention.
Appropriateness of eligibility criteria, baseline and outcome measures, recording of sessions, and randomisation protocol. | From the date of randomisation to date of final follow-up, up to 1 year.
  Rates of enrolment and drop out will be recorded. Fidelity of the intervention will be assessed by video recording.
Estimating sample size needed for Phase III RCT. | From the start of the data analysis to study completion date, up to 6 months.
  Sample size calculations will be conducted during the primary analysis.
Completion rates of outcome measures. | 6 months.
  Based on how many participants complete all of the outcome measures.

SECONDARY OUTCOMES:
Multiple Sclerosis Impact Scale-29 | Baseline, 3-months post randomisation, 6-month post randomisation
  Non-cognitive questionnaire; Reliable Change Index between groups. Scores range from 9 to 36. Higher scores indicate greater psychological impact of MS on everyday life.
Everyday Memory Questionnaire-participant. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Cognitive questionnaire; Reliable Change Index between groups. Scores range from 0 to 112. Higher scores indicate more frequent memory problems.
Everyday Memory Questionnaire-relative. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Cognitive questionnaire; Reliable Change Index between groups. Scores range from 0 to 112. Higher scores indicate more frequent memory problems.
General Health Questionnaire-30. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Non-cognitive questionnaire; Reliable Change Index between groups. Scores range from 0 to 90. Higher scores indicate increased psychological distress.
Fatigue Severity Scale. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Non-cognitive questionnaire; Reliable Change Index between groups. Scores range from -3.4 to 3.4. Higher scores indicate a greater impact of fatigue.
EuroQol-5 Dimensions, five-level version. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Non-cognitive questionnaire; Reliable Change Index between groups. Scores from 0 to 100. Higher scores indicate better overall health.
Guy's Neurological Disability Scale. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Non-cognitive questionnaire; Reliable Change Index between groups. Scores range from 0 to 55. Higher scores indicate increased disability.
Brief Repeatable Battery of Neuropsychological Tests. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Cognitive test; Reliable Change Index between groups. Scores ranges vary depending on the individual test. Higher scores indicate better performance.
Doors and People test. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Cognitive test; Reliable Change Index between groups. Scores range from 0 to 20. Higher scores indicate better performance.
Trail Making Test. | Baseline, 3-months post randomisation, 6-month post randomisation.
  Cognitive test; Reliable Change Index between groups. Scores range from 0 to 20. Higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Roshan das Nair, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom